CLINICAL TRIAL: NCT03545321
Title: Intervention to Increase Naloxone Engagement and Distribution in Community Pharmacies: A Four-State Randomized Trial
Brief Title: RESPOND TO PREVENT: Stepwise Pharmacy Naloxone Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brandeis University (Other)
Collaborators: Comagine Health (Other); Oregon Health and Science University (Other); University of Rhode Island (Other); University of Washington (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-37685; R01DA045745 (NIH)
Record Dates: First submitted 2018-05-08; First posted 2018-06-04 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Pharmacies; Opioid Use; Patient Safety
Keywords: Naloxone; Community pharmacies; Academic detailing; MOON; MOON+; RESPOND
MeSH Terms: interventions — Moon

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOON+ (Experimental): MOON+ includes pharmacist online training on opioid safety and naloxone provision, academic detailing of the pharmacy, materials for use at the pharmacy, standardized overdose response safety protocols, and reminder tools for training reinforcement
  Interventions: Behavioral: MOON+

INTERVENTIONS:
Behavioral: MOON+ — MOON+ is an intervention to support the pharmacy and pharmacist to improve opioid safety and naloxone provision. Materials include educational trainings, materials for use with pharmacists, information for patients, and materials for standardizing overdose safety at the pharmacy

SUMMARY:
This multi-site study will test the efficacy of an intervention to train and equip pharmacists to provide naloxone, an overdose antidote, to patients using prescribed and illicit opioids, to improve opioid safety and prevent opioid-involved adverse events. The study will carry out a stepped-wedge, cluster randomized trial implemented over five waves, within two chain community pharmacies across four states with varying pharmacy-based naloxone distribution laws: Oregon, Washington, Massachusetts, and New Hampshire. Our specific study aims are to: 1) integrate two successful demonstration research projects into one cohesive educational program (MOON+), 2) evaluate the effectiveness of MOON + on naloxone-related outcomes, and 3) use mixed methods to further explore the impact and implementation of MOON+ and associated factors (e.g., state policy, store policy, region).

DETAILED DESCRIPTION:
The purpose of this study is to integrate two pharmacy-focused educational interventions designed to increase pharmacy based naloxone (PBN) dispensing and improve opioid safety. The intervention is comprised of two successful demonstration research projects (RESPOND, PI: Hartung; MOON, PI: Green), which include online and one-on-one educational outreach (i.e. academic detailing) demonstrated to provide knowledge and training for pharmacists to identify and effectively engage with patients who may be at high-risk for an opioid overdose. This study tests the combined interventions' effectiveness at improving opioid safety engagement and naloxone-related outcomes in community pharmacies. The following primary specific aims will drive this research:

For Aim 1: The research team and study pharmacy partners will work collaboratively to integrate MOON and RESPOND into MOON+, including the creation of a website to host intervention components. Feedback from community partners and pharmacy professional associations will be sought to finalize the MOON+ content and materials.

For Aim 2: We will conduct a stepped wedge, cluster randomized design in 160 pharmacies throughout Oregon, Washington, Massachusetts, and New Hampshire. Implementation will occur across five waves, each of which will include a baseline survey, toolkit orientation session, academic detailing, an online course, and access to printed onsite materials (algorithm, checklists, stickers, posters). The targeted population is pharmacists and pharmacy managers in CVS pharmacies (MA and NH) and Albertsons Companies (OR and WA) across the study states and who volunteer to participate in the educational intervention. We will recruit 40 pharmacies per state, 160 pharmacies total, providing a sample of approximately 450 pharmacist participants. Each store will have a pharmacy champion (a pharmacist or pharmacy manager), who will be the point of contact for the intervention. Only pharmacies with a consenting pharmacy champion will be eligible for the study; pharmacists at those sites may opt to participate. Data collection will occur at baseline, 6-, and 12-month follow-up, using surveys (pharmacist-level), store dispensing data and daily faxed counts of naloxone encounters (store-level). Note that no identifiable health information about the patients will be collected in these forms, only basic counts and communication descriptors. The follow up surveys for pharmacists consist of brief questionnaires about the training, attitudes and perceptions of naloxone and naloxone dispensing, sale of syringes over the counter, and dispensing of buprenorphine.

For Aim 3: We will use a mixed methods approach to identify facilitators and barriers (e.g. state-specific policies, store policies, region) to intervention implementation and effectiveness. Methods will include an environmental scan of extant laws and policies, fidelity checking, pharmacist focus groups (n=50), and interviews with patients who have received or would be eligible for receiving naloxone (n=28).

ELIGIBILITY:
Inclusion Criteria:

* English speaking, age 18 years or older, a pharmacist or pharmacy manager employed half time or more by CVS Pharmacy in Massachusetts or New Hampshire or by Albertsons Companies in Washington or Oregon

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
6 month change in naloxone distribution rates from study pharmacies | baseline, six months post intervention
  Naloxone fill data from study pharmacies
12 month change in naloxone distribution rates from study pharmacies | baseline, 12 months post intervention
  Naloxone fill data from study pharmacies
6 month change in naloxone-related patient engagement in the pharmacy | baseline, six months post intervention
  counts of naloxone-related conversations between pharmacy staff and patients and friends/family of opioid users will be recorded in a MOON+ log book by pharmacy staff
12 month change in naloxone-related patient engagement in the pharmacy | baseline, 12 months post intervention
  counts of naloxone-related conversations between pharmacy staff and patients and friends/family of opioid users will be recorded in a MOON+ log book by pharmacy staff

SECONDARY OUTCOMES:
baseline pharmacist self-reported changes | baseline
  A 73 item questionnaire developed by the investigators will be used to collect data on knowledge, attitudes, perceived behavioral control, and self-efficacy toward dispensing naloxone. It has 5 sections: demographics (8 questions), experience within the pharmacy setting (18 questions), knowledge and experience with naloxone (19 questions), experience with overdose response (10 questions), overdose prevention and use of naloxone scenarios (18 questions). The questions use both multiple choice and likert scales formats.
6 month pharmacist self-reported changes | six months post intervention
  A 73 item questionnaire developed by the investigators will be used to collect data on knowledge, attitudes, perceived behavioral control, and self-efficacy toward dispensing naloxone. It has 5 sections: demographics (8 questions), experience within the pharmacy setting (18 questions), knowledge and experience with naloxone (19 questions), experience with overdose response (10 questions), overdose prevention and use of naloxone scenarios (18 questions). The questions use both multiple choice and likert scales formats.
12 months pharmacist self-reported changes | 12 months post intervention
  A 73 item questionnaire developed by the investigators will be used to collect data on knowledge, attitudes, perceived behavioral control, and self-efficacy toward dispensing naloxone. It has 5 sections: demographics (8 questions), experience within the pharmacy setting (18 questions), knowledge and experience with naloxone (19 questions), experience with overdose response (10 questions), overdose prevention and use of naloxone scenarios (18 questions). The questions use both multiple choice and likert scales formats.

CONTACTS AND LOCATIONS:
Overall Officials: Traci C Green, PhD, MSc, Principal Investigator — Brandeis University
Locations (5):
- United States (5):
  - Brandeis University, Waltham, Massachusetts
  - Comagine Health, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Rhode Island, Kingston, Rhode Island
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data will be shared with other researchers upon request.

REFERENCES:
- [Derived] Blough MJ, Rocha A, Bratberg J, Silcox J, Bolivar D, Floyd AS, Gray M, Green TC. The Cost of Safe Injection: Insights on Nonprescription Syringe Price Variability From Systematic Secret Shopping. Subst Use Addctn J. 2024 Apr;45(2):201-210. doi: 10.1177/29767342231217831. Epub 2024 Jan 4. PMID 38258818
- [Derived] Green TC, Silcox J, Bolivar D, Gray M, Floyd AS, Irwin AN, Hansen RN, Hartung DM, Bratberg J. Pharmacy staff-reported adaptations to naloxone provision and over-the-counter (OTC) syringe sales during the COVID-19 pandemic: Experiences across multiple states and 2 pharmacy chains. J Am Pharm Assoc (2003). 2024 Jan-Feb;64(1):71-78. doi: 10.1016/j.japh.2023.10.014. Epub 2023 Oct 18. PMID 37863398